CLINICAL TRIAL: NCT04971356
Title: Aspirin Plus Ticagrelor for 1 Month Followed by 5 Months Ticagrelor Monotherapy Versus Aspirin Plus Ticagrelor for 12 Months in Acute Coronary Syndrome Patients With Drug-coated Balloon: a Multicentre, Randomized, Non-inferiority Trial
Brief Title: 1-month DAPT Plus 5-month Ticagrelor Monotherapy Versus 12-month DAPT in Patients With Drug-coated Balloon
Acronym: CAGEFREEII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, LingTao, Professor in cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAGE-FREE II
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Antiplatelet Drug; Acute Coronary Syndrome; Angioplasty, Balloon
Keywords: Ticagrelor Monotherapy; Acute coronary syndrome; Drug-coated balloons
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): 1-month of Aspirin + Ticagrelor, followed by 5-month of Ticagrelor monotherapy; Afterward, Aspirin monotherapy for 6 months
  Interventions: Drug: Aspirin 100mg for 1-month (immediately after PCI); Drug: Ticagrelor 90mg for 6-month (immediately after PCI); Drug: Aspirin 100mg for 6-month (6-month post PCI)
- Reference arm (Active Comparator): 12-month Aspirin plus Ticagrelor
  Interventions: Drug: Aspirin 100mg for 12-month (immediately after PCI); Drug: Ticagrelor 90mg for 12-month (immediately after PCI)

INTERVENTIONS:
Drug: Aspirin 100mg for 1-month (immediately after PCI) — Aspirin for 1-month immediately after PCI to be a part of medication treatment in the Experimental arm
  Arms: Experimental arm
Drug: Ticagrelor 90mg for 6-month (immediately after PCI) — Ticagrelor for 6-month immediately after PCI to be a part of medication treatment in the Experimental arm
  Arms: Experimental arm
Drug: Aspirin 100mg for 6-month (6-month post PCI) — Aspirin for 6-month at 6 months post-PCI (after the discontinuation of the 6-month Ticagrelor treatment) to be a part of medication treatment in the Experimental arm
  Arms: Experimental arm
Drug: Aspirin 100mg for 12-month (immediately after PCI) — Aspirin for 12-month immediately after PCI to be a part of medication treatment in the Reference arm
  Arms: Reference arm
Drug: Ticagrelor 90mg for 12-month (immediately after PCI) — Ticagrelor for 12-month immediately after PCI to be a part of medication treatment in the Reference arm
  Arms: Reference arm

SUMMARY:
Drug-Coated Balloon (DCB) angioplasty is similar to plain old balloon angioplasty procedurally, but there is an anti-proliferative medication paclitaxel coated to the balloon. Treating ISR lesions with the DCB has the theoretical advantage of avoiding multiple stent layers and respecting the vessel anatomy. DCB has shown promising results for the treatment of ISR. Currently, DCB has a Class I indication to treat ISR recommended by European Society of Cardiology guidelines. In addition, some interventional cardiologist has also applied DCB in de novo lesions in their clinical practice.

Bleeding after PCI remains a substantial clinical problem. Bleeding post-PCI increases the risk of adverse outcomes such as death, non-fatal myocardial infarction, and prolongs hospital stay. Clinical data has suggested that major bleeding post-PCI would increase the risk of mortality 5.7-fold. The antiplatelet medications are the major cause of bleeding events post-PCI.

Current guidelines for stents recommended DAPT of aspirin plus a P2Y12 inhibitor for at least 12 months after stent implantation in patients with the acute coronary syndrome. Compared with the DES, because of the absence of metal inside the coronary artery, the use of DCB might theoretically allow shorter duration antiplatelet therapy. However, the optimal course of DAPT for the DCB treated patients remains controversial.

In 2013, the consensus from the German group suggested that for the acute coronary syndrome, DAPT should be used for 12 months. The consensus of DAPT developed by the European Society of Cardiology (ESC) in 2017 stated that "in patients treated with DCB, dedicated clinical trials investigating the optimal duration of DAPT are lacking." So far, there are no randomized data showing the optimal DAPT duration for the DCB treated patients.

In the current study, we use Aspirin + Ticagrelor for 1-month followed by Ticagrelor monotherapy for 5-month, afterward, Aspirin monotherapy for 6 months to be the antiplatelet regimen in the experimental arm, to compare with the Reference arm, which is Aspirin + Ticagrelor for 12-month in a non-inferiority statistical assumption, aiming to investigate the optimal duration of the DAPT in ACS patients after DCB treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an indication for PCI due to acute coronary syndrome
2. All target lesions can be successful treatment of PCI with drug-coated balloon (DCB)
3. Patients who are able to complete the follow-up and compliant to the prescribed medication

Exclusion Criteria:

1. Under the age of 18 or Older than 80 years old
2. Unable to give informed consent
3. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
4. Known contraindication to medications such as Heparin, antiplatelet drugs, or contrast.
5. Currently participating in another trial and not yet at its primary endpoint
6. Planned elective surgery
7. Concurrent medical condition with a life expectancy of less than 1 years
8. Previous intracranial haemorrhage
9. Need long-term oral anticoagulant therapy
10. Cardiogenic shock
11. Previous stent implantation 6 month
12. In-stent thrombosis
13. Target lesion located in surgical conduit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1948 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 12 months
  NACE is a composite clinical endpoint of all-cause death, any stroke, any MI, any revascularization and BARC type 3 or 5 bleeding events

SECONDARY OUTCOMES:
Any ischemic or bleeding event | 1, 6 and 12 months
  Any ischemic and bleeding event includes any all-cause death, any stroke, MI, BARC-defined type 3 bleeding, any revascularization and BARC-defined type 2 bleeding events
BARC type 3 or 5 bleeding events | 1, 6 and 12 months
  Bleeding events type 3 or 5 defined by BARC (Bleeding Academic Research Consortium) criteria
BARC type 2 ,3 or 5 bleeding events | 1, 6 and 12 months
  Bleeding events type 2, 3 or 5 defined by BARC (Bleeding Academic Research Consortium) criteria
BARC defined type 2 bleeding events | 1, 6 and 12 months
  Bleeding events type 2 defined by BARC (Bleeding Academic Research Consortium) criteria
Rate of NACE | 1 and 6 months
  NACE is a composite clinical endpoint of all-cause death, any stroke, any MI, any revascularization and BARC type 3 or 5 bleeding events
Device-oriented Composite Endpoint (DoCE) | 1, 6 and 12 months
  DoCE is a composite clinical endpoint of cardiac cause death, target vessel myocardial infraction (TV-MI), and Clinically individual target lesion revascularization (CI-TLR)
Cardiac death | 1, 6 and 12 months
  Rates of individual components of DoCE
Target vessel myocardial infraction (TV-MI) | 1, 6 and 12 months
  Rates of individual components of DoCE
Clinically individual target lesion revascularization (CI-TLR) | 1, 6 and 12 months
  Rates of individual components of DoCE
Patient-oriented Composite Endpoint (PoCE) | 1, 6 and 12 months
  The primary safety endpoint of PoCE is defined as all-cause death, any stroke, any MI, any revascularization
All-cause death | 1, 6 and 12 months
  Rates of individual components of PoCE
Any MI | 1, 6 and 12 months
  Rates of individual components of PoCE
Any stroke | 1, 6 and 12 months
  Rates of individual components of PoCE
Any revascularization | 1, 6 and 12 months
  Rates of individual components of PoCE
Target vessel failure (TVF) | 1, 6 and 12 months
  Target vessel failure is defined as cardiovascular death, target vessel myocardial infraction (TV-MI), and clinically-indicated target vessel revascularization
Clinically-indicated target vessel revascularization | 1, 6 and 12 months
  Rates of individual components of TVF
Definite/Probable stent thrombosis rates | 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD,PHD, Study Chair — Xijing Hospital; Patrick Serruys, MD,PHD, Study Chair — National University of Ireland, Galway; Yoshinobu Onuma, MD,PHD, Study Chair — National University of Ireland, Galway; Chao Gao, MD,PHD, Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao C, Zhu B, Ouyang F, Wen S, Xu Y, Jia W, Yang P, He Y, Zhong Y, Zhou Y, Guo Z, Shen G, Ma L, Xu L, Xue Y, Hu T, Wang Q, Liu Y, Zhang R, Liu J, Jiang Z, Xia J, Garg S, van Geuns RJ, Capodanno D, Onuma Y, Wang D, Serruys P, Tao L; REC-CAGEFREE II Investigators. Stepwise dual antiplatelet therapy de-escalation in patients after drug coated balloon angioplasty (REC-CAGEFREE II): multicentre, randomised, open label, assessor blind, non-inferiority trial. BMJ. 2025 Mar 31;388:e082945. doi: 10.1136/bmj-2024-082945. PMID 40164448
- [Derived] Gao C, Zhu B, Liu J, Jiang Z, Hu T, Wang Q, Liu Y, Yuan M, Li F, Zhang R, Xia J, Onuma Y, Wang D, Serruys P, Tao L; REC-CAGEFREE II Study Group. Randomized evaluation of 5-month Ticagrelor monotherapy after 1-month dual-antiplatelet therapy in patients with acute coronary syndrome treated with drug-coated balloons: REC-CAGEFREE II trial rationale and design. BMC Cardiovasc Disord. 2024 Jan 20;24(1):62. doi: 10.1186/s12872-024-03709-1. PMID 38245724